CLINICAL TRIAL: NCT04735315
Title: Assessment of Renal Function in Adults Born Preterm: The HAPI-Kidney Study
Status: Active, not recruiting | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); European Georges Pompidou Hospital (Other); Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Anne Monique NUYT,MD, Chair and Chief, Department of Pediatrics, Faculty of Medicine University of Montreal / CHU Sainte-Justine, St. Justine's Hospital
Other Study IDs: HAPI-Kidneys
Record Dates: First submitted 2021-01-14; First posted 2021-02-03 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Prematurity; Extreme
Keywords: Extremely preterm; Clinical study; Developmental origin of adult health and disease; Prematurity; Renal system; Cardiovascular system
MeSH Terms: conditions — Premature Birth; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The team collected the blood and urine of the participants. They kept whole blood and urine the the biobank. The group also isolated the plasma and serum to perform assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Born preterm: Inclusion :
  Born preterm ≤29 weeks Aged 18-40 years Participants with type-2 diabetes
  Exclusion :
  Currently pregnant due to administration of radionucleotides and impact on GFR Severe neurosensory deficit preventing test completion History of characterized kidney disease independent of preterm birth, including type-1 diabetes, glomerulopathies (e.g. nephrotic syndrome, glomerulonephritis), polycystic kidney disease, polycystosis, severe uropathy (Grade 4 or 5 RVU, severe hydronephrosis (SFU IV and V), posterior valve history), history of nephrectomy, exposure to radiotherapy or chemotherapy - given that we are interested in isolating the effects of preterm birth and that prevalence of these conditions is not increased in individuals born preterm In case of contra-indication to MRI scanning (which should be rare in the young population studied), the participant will still be given the opportunity to complete the other examinations.
  Interventions: Other: Preterm birth
- Born term: Inclusion :
  Born full-term at 37-41 weeks Birthweight ˃2500g Aged 18-40 years Participants with type-2 diabetes
  Exclusion :
  Currently pregnant due to administration of radionucleotides and impact on GFR Severe neurosensory deficit preventing test completion History of characterized kidney disease independent of preterm birth, including type-1 diabetes, glomerulopathies (e.g. nephrotic syndrome, glomerulonephritis), polycystic kidney disease, polycystosis, severe uropathy (Grade 4 or 5 RVU, severe hydronephrosis (SFU IV and V), posterior valve history), history of nephrectomy, exposure to radiotherapy or chemotherapy - given that we are interested in isolating the effects of preterm birth and that prevalence of these conditions is not increased in individuals born preterm In case of contra-indication to MRI scanning (which should be rare in the young population studied), the participant will still be given the opportunity to complete the other examinations.
  Interventions: Other: Preterm birth

INTERVENTIONS:
Other: Preterm birth — The study compares young adult subjects born premature (< 29 weeks) versus term > 37-41 weeks)

SUMMARY:
Every year in Canada, 1500 babies are born ≤29 weeks' gestational age (GA) and the majority survive to adulthood. Preterm birth occurs during a critical period of nephrogenesis. Antenatal and postnatal exposure to various insults may permanently disrupt normal kidney development. Indeed, preterm children have reduced nephron number and altered glomerular architecture, which may lead to glomerular hyperfiltration thus perpetuating renal damage. However, the long-term consequences of preterm birth on renal function remain under-studied. The existing reports on glomerular function have yielded contradictory results and were limited by use of imprecise estimates of glomerular filtration rate (GFR) or small sample size. Yet, a registry-based study has shown the increased risk of chronic kidney diseases (CKD) in individuals born preterm.

In addition, individuals born preterm have higher blood pressure. As mechanisms for hypertension following preterm birth are being unravelled, the role of the kidneys, which is key in chronic hypertension, is to be determined. So far, we have shown a relationship between smaller kidney size and increased blood pressure. A better understanding of the early markers of kidney dysfunction following preterm birth will facilitate screening and intervention to halt progression to CKD as there are currently no long-term renal follow-up guidelines for individuals born preterm.

This proposal builds on our previous works on long-term health outcomes of preterm birth and experimental model of prematurity-related conditions and renal development. We aim to assess glomerular function and renal vasoactive regulatory factors in relation to blood pressure using precise measures in a cohort of young adults born preterm ≤29 weeks versus full-term controls. We further take advantage of our previous assessment of this cohort (Health of Adults born Preterm Investigation (HAPI) - CIHR 2014-18) to evaluate changes in estimated GFR and albuminuria over a 5-year period.

DETAILED DESCRIPTION:
Given that preterm birth is associated with reduced nephron endowment and higher glomerular area on renal histology suggesting compensatory glomerular hyperfiltration, we postulate that :

Hypothesis 1: mGFR relative to total kidney volume is higher in adults born preterm vs. to full-term controls.

Hypothesis 2: mGFR relative to kidney volume is associated with plasma renin activity, aldosterone, copeptin and apelin levels. Levels of these vasoactive factors may correlate to blood pressure values.

Hypothesis 3: Rates of decline in eGFR and increase in albuminuria is more important in the preterm vs. full-term group. Hypertension at baseline predicts faster decline in eGFR and increase in albuminuria. Decrease in eGFR and increase in albuminuria correlate with increasing blood pressure over time.

Hypothesis 4: Higher baseline copeptin levels and, reciprocally, lower baseline apelin levels are associated with faster decline in eGFR and increase in albuminuria.

Our overarching aim is to assess long-term glomerular function in adults born preterm ≤29 weeks' GA versus full-term controls.

1. To assess the association between preterm birth and measured GFR, compared to estimated GFR, in young adulthood (18-40 years).
2. To examine the association between mGFR and vasoactive humoral factors involved in kidney hemodynamics (plasma renin activity, aldosterone, copeptin, apelin) in relation to blood pressure in young adults born preterm versus full-term controls.
3. To compare changes in eGFR and albuminuria over a 5-year period in relation to change in blood pressure in young adults born preterm versus full-term controls.
4. To determine whether baseline levels of copeptin and apelin can predict changes in eGFR and albuminuria over a 5-year period in young adults born preterm versus full-term controls.

ELIGIBILITY:
Inclusion Criteria:

* Born preterm ≤29 weeks or full-term at 37-41 weeks;
* For full-term controls only, birthweight ˃2500g;
* Aged 18-40 years;
* Participants with type-2 diabetes can be included.

Exclusion Criteria:

* Currently pregnant due to administration of radionucleotides and impact on GRF,
* Severe neurosensory deficit preventing test completion,
* History of characterized kidney disease independent of preterm birth, including type-1 diabetes, glomerulopathies (e.g. nephrotic syndrome, glomerulonephritis), polycystic kidney disease, polycystosis, severe uropathy (Grade 4 or 5 RVU, severe hydronephrosis (SFU IV and V), posterior valve history), history of nephrectomy, exposure to radiotherapy or chemotherapy - given that we are interested in isolating the effects of preterm birth and that prevalence of these conditions is not increased in individuals born preterm,
* In case of contra-indication to MRI scanning (which should be rare in the young population studied), the participant will still be given the opportunity to complete the other examinations.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are recruited from the HAPI study, which included 101 individuals born ≤29 weeks in the province of Quebec in 1987-97 (including 83 from CHU Ste-Justine (CHUSJ) who were similar to non-participant survivors for neonatal characteristics), and 105 individuals born full-term recruited among friends/siblings and through advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
mGFR relative to kidney volume (scintigraphy), measurement 1 | 90 minutes
  First, whole-kidney mGFR is measured from the plasma clearance of a radionuclide labeled tracer, 99mTc-DTPA, using the slope-intercept method and single-compartment simplification. A single bolus of 300 microcuries (11.1 mega-Becquerels) of 99mTc-DTPA is injected in one arm and plasma sampling for activity concentration (Hidex Automatic Gamma Counter) is performed in the other arm at 90, 120, 150 and 180 minutes. Calculation of mGFR is as follow: mGFR = (Q/Co) x (0.693/T1/2) where Q the injected dose and Co the extrapolated plasmatic activity at time 0.107 If needed, correction for the rapid component of the time activity curve is performed using the Brochner-Mortensen equation. Value of mGFR is then corrected to the patient's BSA, derived from measured weight and height using DuBois' formula, and expressed in mL/min/1.73 m2. Estimated effective dose of the procedure is 0.054 mSv.
mGFR relative to kidney volume (scintigraphy), measurement 2 | 120 minutes
  First, whole-kidney mGFR is measured from the plasma clearance of a radionuclide labeled tracer, 99mTc-DTPA, using the slope-intercept method and single-compartment simplification. A single bolus of 300 microcuries (11.1 mega-Becquerels) of 99mTc-DTPA is injected in one arm and plasma sampling for activity concentration (Hidex Automatic Gamma Counter) is performed in the other arm at 90, 120, 150 and 180 minutes. Calculation of mGFR is as follow: mGFR = (Q/Co) x (0.693/T1/2) where Q the injected dose and Co the extrapolated plasmatic activity at time 0.107 If needed, correction for the rapid component of the time activity curve is performed using the Brochner-Mortensen equation. Value of mGFR is then corrected to the patient's BSA, derived from measured weight and height using DuBois' formula, and expressed in mL/min/1.73 m2. Estimated effective dose of the procedure is 0.054 mSv.
mGFR relative to kidney volume (scintigraphy), measurement 3 | 150 minutes
  First, whole-kidney mGFR is measured from the plasma clearance of a radionuclide labeled tracer, 99mTc-DTPA, using the slope-intercept method and single-compartment simplification. A single bolus of 300 microcuries (11.1 mega-Becquerels) of 99mTc-DTPA is injected in one arm and plasma sampling for activity concentration (Hidex Automatic Gamma Counter) is performed in the other arm at 90, 120, 150 and 180 minutes. Calculation of mGFR is as follow: mGFR = (Q/Co) x (0.693/T1/2) where Q the injected dose and Co the extrapolated plasmatic activity at time 0.107 If needed, correction for the rapid component of the time activity curve is performed using the Brochner-Mortensen equation. Value of mGFR is then corrected to the patient's BSA, derived from measured weight and height using DuBois' formula, and expressed in mL/min/1.73 m2. Estimated effective dose of the procedure is 0.054 mSv.
mGFR relative to kidney volume (scintigraphy), measurement 4 | 180 minutes
  First, whole-kidney mGFR is measured from the plasma clearance of a radionuclide labeled tracer, 99mTc-DTPA, using the slope-intercept method and single-compartment simplification. A single bolus of 300 microcuries (11.1 mega-Becquerels) of 99mTc-DTPA is injected in one arm and plasma sampling for activity concentration (Hidex Automatic Gamma Counter) is performed in the other arm at 90, 120, 150 and 180 minutes. Calculation of mGFR is as follow: mGFR = (Q/Co) x (0.693/T1/2) where Q the injected dose and Co the extrapolated plasmatic activity at time 0.107 If needed, correction for the rapid component of the time activity curve is performed using the Brochner-Mortensen equation. Value of mGFR is then corrected to the patient's BSA, derived from measured weight and height using DuBois' formula, and expressed in mL/min/1.73 m2. Estimated effective dose of the procedure is 0.054 mSv.
Whole-kidney GFR (MRI) | 1 hour
  Whole-kidney GFR is a product of nephron number and single-nephron GFR. As a surrogate for single-nephron GFR, we are examining mGFR in relation to total kidney volume (i.e. mGFR per cm3 of kidney volume), which is reduced in adults born preterm and correlates to a certain extent to nephron number. Total kidney volume is measured by multi-parametric magnetic resonance imaging (MRI), which also allows for a comprehensive assessment of kidney structure and hemodynamics. No contrast is injected. Images are acquired using a Philips Ingenia 1.5T MRI system and a 16/32 channels dStream Torso coil (Philips). To quantify total kidney volume, localizer scans at end expiration are acquired using balanced turbo field echo and balanced fast field echo in three orthogonal planes. Volume is then calculated by manually tracing the kidney on the coronal images using Philips Intellispace Portal.
Rate of glomerular hyperfiltration | 30 minutes
  We also examine rate of glomerular hyperfiltration, which is typically described as ˃95th percentile of a reference population. The prevalence of single-nephron glomerular hyperfiltration is estimated by assessing the proportion of participants born preterm with a ratio of mGFR to total kidney volume ˃95th percentile calculated in participants born full-term.

SECONDARY OUTCOMES:
Biomarker of vasoregulatory mechanisms, kidney level, Renin | 60 minutes
  Plasma renin activity is determined by measuring the mass of angiotensin-1 generated per volume of human plasma in one hour, using a PRA ELISA assay (IBL-America, MN, USA).
Biomarker of vasoregulatory mechanisms, kidney level, Aldosterone | 60 minutes
  Plasma aldosterone is assessed using a high sensitivity ELISA assay (IBL-America), with a range of 7.75 - 1000 pg/ml and expected plasma aldosterone values of at least 40 pg/ml113.
Biomarker of vasoregulatory mechanisms, kidney level, Copeptin | 60 minutes
  Plasma copeptin is assessed in the plasma using the BRAHMS KRYPTOR compact PLUS system available at London Health Sciences Centre, London, ON.
Biomarker of vasoregulatory mechanisms, kidney level, Apelin | 60 minutes
  Plasma apelin-12 is assessed using an ELISA assay (Phoenix Pharmaceuticals, CA, USA).
Blood pressure | 10 minutes
  Blood pressure (systolic and diastolic) is measured after seated rest for 5 min before blood sampling using an automated oscillometric device (Dinamap, GE Healthcare) according to the Canadian Hypertension Education Program. Blood pressure is measured in both arms and the average of 3 measures taken at 1-min intervals on the arm with highest readings is used. Participants also undergo 24-hour ambulatory blood pressure measurement (ABPM, Spacelabs Medical, Washington) on their non-dominant arm.
Albuminuria | 5 minutes
  Albumin to creatinine ratio (ACR) is obtained from a spot urine collection.
Estimated GFR | 5 minutes
  Estimated GFR is calculated using validated Full Age Spectrum (FAS) equation, with and without correction for height115 (with IDMS standardized creatinine), as this equation has been shown to be more accurate than the CKD-Epi equation in young adults.
Renal ultrasound and Doppler, Volume | 10 minutes
  Morphologic studies of kidneys including size (volume)
Renal ultrasound and Doppler, Echogenicity | 10 minutes
  Morphologic studies of kidneys including echogenicity (cortex and medulla)
Renal ultrasound and Doppler, urinary tract | 10 minutes
  Morphologic studies of kidneys including urinary tract
Renal ultrasound and Doppler, arterial resistive index | 10 minutes
  Morphologic studies of kidneys including arterial resistive index.
Liver echography | 15 minutes
  Morphologic study of the liver using the echography machine, including the volume.
Muscle ultrasound | 10 minutes
  Ultrasound imaging examinations of the musculoskeletal system, through the rectus femoris muscle. Images of the rectus femoris will be recorded while the participant is in a sitting position.
Muscle elastography | 30 minutes
  For the elastography, the participant will stay still while the share wave is applied. Finally, ultrasound images of the rectus femoris will be recorded in three different states: 1) relaxed position, 2) maximal voluntary contraction and 3) sub-maximal voluntary contraction, using a dynamometer. A 30-second rest period will be implemented between contractions to minimize potential fatigue effects.
Muscular strength | 15 minutes
  Measured in accordance with the standardized test protocol produced by the Canadian Society for Exercise Physiology (CSEP, 2013), using a dynamometer.
Muscular endurance | 15 minutes
  Measured in accordance with the standardized test protocol produced by the Canadian Society for Exercise Physiology (CSEP, 2013), using a dynamometer.
Physical activity | 7 days
  Measured using accelerometry for 7 seven consecutive days.
Aerobic capacity and endurance test | 6 minutes
  Six-minute walking test (6MWT) assesses distance walked over 6 minutes.
Questionnaire #1 | 5 minutes
  Current medication, alcohol, drugs use 2)
Hydration levels, plasma electrolytes | 15 minutes
  Plasma electrolytes measured by the Hospital clinical biochemistry.
Hydration levels, plasma osmolality | 30 minutes
  Plasma osmolality measured by the Hospital clinical biochemistry.
Hydration levels, urine electrolytes | 30 min
  Urine (spot) electrolytes measured by the Hospital clinical biochemistry.
Hydration levels, urine osmolality | 30 minutes
  Urine (spot) osmolality measured by the Hospital clinical biochemistry.
Hydration levels, plasma hematocrit | 30 minutes
  Plasma hematocrit measured by the Hospital clinical biochemistry.
Hydration levels, plasma total proteins | 30 minutes
  Plasma total proteins measured by the Hospital clinical biochemistry.
Cardiometabolic risk factors, glycated hemoglobin | 15 minutes
  Glycated hemoglobin in plasma measured by the Hospital clinical biochemistry.
Cardiometabolic risk factors, plasma lipids | 15 minutes
  Plasma lipids measured by the Hospital clinical biochemistry.
Cardiometabolic risk factors, BMI | 15 minutes
  BMI, calculated using the weight in kg and the height in meters.
Cardiometabolic risk factors, waist-to-hip | 10 minutes
  Waist-to-hip ratio using the measurement of the hip and waist in centimeters
Questionnaire # 2 | 10 minutes
  Socio-economic status from the parents and the participant Occupation and education level (achieved or ongoing), parental education/income for students, primary earner status, personal income. Family history: Parental health history of cardiovascular, metabolic or renal diseases.
Questionnaire #3 | 2 hours
  Obstetrical and neonatal history: (a) maternal: smoking, prepregnancy BMI, hypertension, diabetes, prenatal corticosteroids, chorioamnionitis Neonatal: GA (based on date of last period and/or obstetric ultrasound), birth weight and percentile as per Hadlock for preterm subjects (intrauterine growth curves) and Kramer (postnatal birth weight) for term controls, APGAR, major complications/conditions (mechanical ventilation, O2 and parenteral nutrition duration, umbilical arterial lines, sepsis, acute renal failure, necrotizing enterocolitis, bronchopulmonary dysplasia, ultrasound brain lesions, surgeries, medications (nephrotoxic antibiotics, steroids, indomethacin, diuretics), and length of hospital stay). Data are obtained from medical records.
SF-36 | 10 minutes
  Quality of life and functional status
WHO questionnaire | 10 minutes
  Quality of life and functional status
Diet, food frequency questionnaire | 35 minutes
  Food frequency questionnaire
Diet, 24-hour meal interview | 10 minutes
  24-hour meal interview
MAPA | 24 hours
  Monitoring device for 24 hours blood pressure measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Monique Nuyt, MD, Principal Investigator — StJustine's Hospital; Thuy Mai Luu, MD, Principal Investigator — StJustine's Hospital
Locations (1):
- StJustine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: 1 year after all the results are published
Access Criteria: Request of collaboration through data access will be examined by the PI's.